CLINICAL TRIAL: NCT06439342
Title: An Open-label, Single-arm Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of Maribavir in Chinese Transplant Recipients With Cytomegalovirus (CMV) Infections That Are Refractory or Resistant to Treatment With Ganciclovir, Valganciclovir, Cidofovir or Foscarnet
Brief Title: A Study of Maribavir in Chinese Adults With Cytomegalovirus (CMV) Infections
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-620-3002
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Cytomegalovirus (CMV)
MeSH Terms: interventions — maribavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maribavir (Experimental): Participants will receive maribavir 400 milligrams (mg), tablets, orally twice a day (BID) for up to 8 weeks.
  Interventions: Drug: Maribavir

INTERVENTIONS:
Drug: Maribavir — Maribavir tablets
  Other Names: TAK-620

SUMMARY:
The main aim of this study is to learn how safe maribavir is in Chinese adults who have undergone hematopoietic stem cell or organ transplantation and have a cytomegalovirus (CMV) infection and how well they tolerate treatment with maribavir. Other aims are to see how effective maribavir is in treating CMV infection and getting rid of the symptoms, the recurrence rate of CMV infection after treatment with maribavir and if the treatment is required again. Researchers will also check for changes (mutations) occurring in the virus which may cause treatment with maribavir to no longer work well or to not work at all (resistance to maribavir).

The participants will be treated with maribavir for 8 weeks.

During the study, participants will visit their study clinic 18 times.

ELIGIBILITY:
Inclusion Criteria

* The participant or the participant's legally acceptable representative is willing and able to understand and fully comply with study procedures and requirements, in the opinion of the investigator.
* The participant/participant's legally representative has provided informed consent (that is, in writing, documented via a signed and dated informed consent form [ICF]) and any required privacy authorization prior to the initiation of any study procedures.
* The participant is aged 18 years or older (ie, greater than or equal to [>=] 18 years) at the time of signing the ICF.
* The participant must be of Chinese descent, defined as born in China and having Chinese parents and Chinese maternal and paternal grandparents.
* The participant must be a recipient of hematopoietic stem cell or solid organ transplant.
* The participant must have a documented CMV infection in whole blood or plasma, with a screening value of >=1,365 International unit per milliliter IU/mL in whole blood or >=455 IU/mL in plasma in 2 consecutive assessments, separated by at least 1 day, as determined by local laboratory quantitative polymerase chain reaction (qPCR) or comparable quantitative CMV DNA results. Both samples should be taken within 14 days prior to receiving the investigational product with second sample obtained within 5 days prior to receiving the investigational product. The same laboratory and same sample type (whole blood or plasma) must be used for these assessments.
* The participant must have a current CMV infection that is refractory to the most recently administered of the 4 anti-CMV treatment agent(s) eg, intravenous (IV) ganciclovir/oral valganciclovir, IV foscarnet, or IV cidofovir. Refractory is defined as documented failure to achieve greater than (>) 1 log10 (common logarithm to base 10) decrease in CMV DNA level in whole blood or plasma after a 14 day or longer treatment period with the above 4 agents.
* Participants who have documentation of 1 or more CMV genetic mutations associated with resistance to ganciclovir/valganciclovir, cidofovir, or foscarnet must also meet the definition of refractory CMV infection.
* Have all the following results as part of screening laboratory assessments:

  * Absolute neutrophil count >=1000 per cubic millimeter (/mm^3) (1*10^9 per liter [/L]).
  * Platelet count >= 25,000/mm^3 (25*10^9/L)
  * Hemoglobin >= 8 grams per deciliter (g/dL)
  * Estimated glomerular filtration rate >= 30 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) as assessed by Modification of Diet in Renal Disease (MDRD) formula.
* The participant must have life expectancy of at least 8 weeks.
* The participant has a body weight of at least 35 kilogram (kg).
* The female participant either be of nonchildbearing potential, or if of childbearing potential then have a negative serum human chorionic gonadotropin (hCG) or beta-hCG (β-hCG) pregnancy test at screening. Males, or nonpregnant, nonlactating female participants who are sexually active must agree to comply with the applicable contraceptive requirements of this protocol during the investigational product administration period and for 90 days after the last dose of investigational product.
* The participant must be able to swallow tablets, or receive tablets crushed and/or dispersed in water via a nasogastric or orogastric tube.

Exclusion Criteria:

* The participant has CMV disease with central nervous system (CNS involvement) (eg, CMV encephalitis) or ophthalmic involvement (eg, CMV retinitis) as assessed by the investigator at the time of screening.
* That participant has uncontrolled other type of infection as assessed by the investigator on the date of treatment assignment.
* The participant has a history of clinically relevant alcohol or drug abuse that may interfere with treatment compliance or assessments with the protocol as determined by the investigator.
* The participant has a known hypersensitivity to maribavir or to any excipients.
* The participant has severe vomiting, diarrhea, or other severe gastrointestinal (GI) illness within 24 hours prior to the first dose of investigational product or a GI absorption abnormality that would preclude administration of oral medication.
* The participant has any clinically significant medical or surgical condition that, in the investigator's opinion, could interfere with interpretation of study results, contraindicate the administration of the investigational product, or compromise the safety or well-being of the participant.
* The participant is receiving valganciclovir, ganciclovir, cidofovir, foscarnet, letermovir, leflunomide, or artesunate when investigational product is initiated, or anticipated to require one of these agents during the 8-week treatment period.
* The participant requires mechanical ventilation or vasopressors for hemodynamic support at the time of baseline.
* The participant has previously received maribavir.
* The participant has previously completed, discontinued, or have been withdrawn from this study.
* The participant has received any investigational agent with known anti-CMV activity within 30 days before initiation of investigational product or CMV vaccine at any time.
* The participant has received any investigational agent or device within 30 days before initiation of investigational product.
* The participant has serum aspartate aminotransferase (AST) >5 times upper limit of normal (ULN) at screening, or serum alanine aminotransferase (ALT) >5 times ULN at screening, or total bilirubin >=3.0 × ULN at screening (except for documented Gilbert's syndrome), by a local laboratory. Note: Participants with biopsy confirmed CMV hepatitis will not be excluded from study participation despite AST or ALT >5 times ULN at screening.
* The participant has known (previously documented) positive results for human immunodeficiency virus (HIV). Participant must have a confirmed negative HIV test result within 3 months of study entry or, if unavailable, be tested by a local laboratory during the screening period.
* The participant has active malignancy with the exception of nonmelanoma skin cancer, as determined by the investigator. Participants who experience relapse or progression of their underlying malignancy (for which hematopoietic stem-cell transplantation (HSCT) or solid organ transplant (SOT) was performed), as determined by the investigator, are not to be enrolled.
* The participant is undergoing treatment for acute or chronic hepatitis C and hepatitis B.
* The participant is pregnant or expecting to conceive or nursing/breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAE), and Adverse Events of Special interest (AESIs) | From first dose of study drug up to Week 20
  TEAEs will be defined as those with a start date on or after the first dose of study treatment, or with a start date before the date of first dose of study treatment but increasing in severity after the first dose of study treatment. An SAE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above-mentioned criteria. AESIs is defined as any adverse event of special interest.
Number of Participants With Clinically Significant Changes in Vital Signs | From first dose of study drug up to Week 20
  Vital signs will include temperature, arterial blood pressure (systolic and diastolic) and pulse. Any change in vital signs assessments which will be deemed clinically significant by the investigator will be reported.
Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters | From first dose of study drug up to Week 20
  Clinical laboratory parameters will include chemistry, hematology, and urinalysis. Any clinical laboratory abnormalities which will be deemed clinically significant by the investigator will be recorded.
Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings | From first dose of study drug up to Week 20
  12-lead ECG will be evaluated. Any ECG assessments which will be deemed clinically significant by the investigator will be reported.
Number of Participants Who will Discontinue From the Study Drug and Study | From first dose of study drug up to Week 20
  Participants discontinuing the study drug treatment and the study will be reported.

SECONDARY OUTCOMES:
Percentage of Participants With Confirmed Clearance of Plasma CMV Deoxyribose Nucleic Acid (DNA) (CMV Viremia Clearance) at Week 8 | At Week 8
  Confirmed CMV viremia clearance is defined as plasma CMV DNA concentration below the lower limit of quantification (<LLOQ), when assessed by CMV Test (Roche COBAS CMV 6800/8800) at a central specialty laboratory, in 2 consecutive postbaseline samples, separated by at least 5 days, regardless of whether either study-assigned treatment was discontinued before the end of the stipulated 8 weeks of therapy.
Percentage of Participants With Achievement of CMV Viremia Clearance and CMV Infection Symptom Control at Weeks 8, 12, 16, and 20 | At Weeks 8, 12, 16 and 20
  Confirmed CMV viremia clearance is defined as plasma CMV DNA concentration below the lower limit of quantification (<LLOQ), when assessed by CMV Test (Roche COBAS CMV 6800/8800) at a central specialty laboratory, in 2 consecutive postbaseline samples, separated by at least 5 days, regardless of whether either study-assigned treatment was discontinued before the end of the stipulated 8 weeks of therapy. Symptom control is defined as resolution or improvement of tissue invasive CMV disease or CMV syndrome for participants symptomatic at baseline or no new symptoms of tissue invasive CMV disease or CMV syndrome for participants asymptomatic at baseline. This outcome measure will be assessed regardless of whether participants complete the stipulated 8 weeks of study-assigned treatment.
Percentage of Participants With Achievement of CMV Viremia Clearance and CMV Infection Symptom Control at Week 8 (After Completion of 8 Weeks Therapy) | At Week 8
  Confirmed CMV viremia clearance will be defined as plasma CMV DNA concentration <LLOQ, when assessed by CMV Test (Roche COBAS CMV 6800/8800) at a central specialty laboratory, in 2 consecutive postbaseline samples, separated by at least 5 days (after completion of 8 weeks therapy). Symptom control is defined as resolution or improvement of tissue invasive CMV disease or CMV syndrome for participants symptomatic at baseline or no new symptoms of tissue invasive CMV disease or CMV syndrome for participants asymptomatic at baseline.
Percentage of Participants With Achievement of CMV Viremia Clearance and CMV Infection Symptom Control After Completion of 8 weeks Therapy Followed by Maintenance of This Treatment Effect Through Weeks 12, 16 and 20 | At Weeks 12, 16 and 20
  Confirmed CMV viremia clearance will be defined as plasma CMV DNA concentration <LLOQ, when assessed by CMV Test (Roche COBAS CMV 6800/8800) at a central specialty laboratory, in 2 consecutive postbaseline samples, separated by at least 5 days (after completion of 8 weeks therapy). Symptom control is defined as resolution or improvement of tissue invasive CMV disease or CMV syndrome for participants symptomatic at baseline or no new symptoms of tissue invasive CMV disease or CMV syndrome for participants asymptomatic at baseline. The maintenance of treatment effect will be based on the achievement of CMV viremia clearance and symptom control at Week 8 after completion of 8 weeks therapy, followed by maintenance of this treatment effect through Weeks 12, 16 and 20.
Percentage of Participants With Recurrence of CMV Viremia During the First 8 Weeks and Through Week 12 to Week 20 | From first dose of study drug up to Week 8, and through Week 12 to Week 20
  Recurrence of CMV viremia is defined as plasma CMV DNA concentrations greater than or equal to (>=) LLOQ, when assessed by central specialty laboratory, in 2 consecutive plasma samples separated by at least 5 days after achieving confirmed viremia clearance.
Percentage of Participants With Recurrence of CMV Viremia During on Treatment and off Treatment | From first dose of study drug up to Week 8 (on treatment) and Week 20 (off treatment)
  Recurrence of CMV viremia is defined as plasma CMV DNA concentrations >= LLOQ, when assessed by central specialty laboratory, in 2 consecutive plasma samples separated by at least 5 days after achieving confirmed viremia clearance. On treatment is the period over which participant received actual dosing (that can be before the stipulated 8 weeks of study-assigned treatment). Off treatment is the period after study treatment.
Percentage of Participants With Recurrence of CMV Viremia Requiring Alternative Treatment After Achieving CMV Viremia Clearance at Study Week 8 | At Week 8
  Recurrence of CMV viremia is defined as plasma CMV DNA concentrations >=LLOQ, when assessed by central specialty laboratory, in 2 consecutive plasma samples separated by at least 5 days after achieving confirmed viremia clearance.
Percentage of Participants With Mutations in the CMV Genes Conferring Resistance to Maribavir | Up to Week 20
  Percentage of participants with mutations in the CMV genes conferring resistance to maribavir will be reported.
Number of Participants With All-cause Mortality During the Study | Up to Week 20
  All-cause mortality during the study will be reported.
Maximum Observed Plasma Concentration (Cmax) at Steady State for Maribavir | Week 1, Day 7: Pre-dose, 0.5, 1.5, 3, 4, 6, 8, and 12 hours post-dose
  Cmax at steady state for maribavir will be assessed.
Time to Reach Cmax (Tmax) at Steady State for Maribavir | Week 1, Day 7: Pre-dose, 0.5, 1.5, 3, 4, 6, 8 and 12 hours post-dose
  Tmax at steady state of maribavir will be assessed.
Minimum Observed Plasma Concentration (Cmin) for Maribavir | Pre-dose and at Weeks 1, 4, and 8
  Cmin of maribavir will be assessed.
Area Under the Plasma Concentration-Time Curve From Time 0 to Time of the Last Quantifiable Concentration Area (AUC0-t) at Steady State for Maribavir | Week 1, Day 7: Pre-dose, 0.5, 1.5, 3, 4, 6, 8 and 12 hours post-dose
  AUC0-t at steady state for maribavir will be assessed.
Area Under the Plasma Concentration-Time Curve Over 1 Dosing Interval of 12 Hours (AUC0-tau) at Steady State for Maribavir | Week 1, Day 7: Pre-dose, 0.5, 1.5, 3, 4, 6, 8 and 12 hours post-dose
  AUC0-tau at steady state for maribavir will be assessed.
Half -life (t1/2) at Steady State for Maribavir | Week 1, Day 7: Pre-dose, 0.5, 1.5, 3, 4, 6, 8 and 12 hours post-dose
  t1/2 at steady state for maribavir will be assessed.
Terminal Elimination Rate Constant (Lambda z) at Steady State for Maribavir | Week 1, Day 7: Pre-dose, 0.5, 1.5, 3, 4, 6, 8 and 12 hours post-dose
  Lambda z at steady state for maribavir will be assessed.
Apparent Volume of Distribution (Vz/F) at Steady State for Maribavir | Week 1, Day 7: Pre-dose, 0.5, 1.5, 3, 4, 6, 8 and 12 hours post-dose
  Vz/F at steady state for maribavir will be assessed.
Apparent Oral Clearance (CL/F) at Steady State for Maribavir | Week 1, Day 7: Pre-dose, 0.5, 1.5, 3, 4, 6, 8 and 12 hours post-dose
  CL/F at steady state for maribavir will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- China (11):
  - Anhui Provincial Hospital(The First Affiliated Hospital of USTC), Hefei, Anhui
  - Xinqiao Hospital Army Medical University, Chongqing, Chongqing Municipality
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Peking University People's Hospital, Beijing, North China
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/912adfb97a4a4dae??page=1&idFilter=TAK-620-3002